CLINICAL TRIAL: NCT01618838
Title: Prospective Endoscopic Safety Evaluation of Late Rectal Mucosal Injury Following CyberKnife Radiosurgery for Clinically Localized Prostate Cancer
Brief Title: Endoscopic Evaluation of Late Rectal Injury Following CyberKnife Radiosurgery for Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study only accrued 4 patients in 2 years, far below target (40). It was closed with no subject reached the primary endpoint, thus no results to publish.
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Sean Collins, M.D., PhD, Assistant Professor, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2009-474
Record Dates: First submitted 2012-06-12; First posted 2012-06-13 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Stage II Prostate Carcinoma
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyberKnife Radiosurgery, Colonoscopy (Other): CyberKnife radiosurgery for prostate cancer; bowel toxicity will be evaluated at 2 years by colonoscopy (lower endoscopy).
  Interventions: Radiation: CyberKnife radiosurgery

INTERVENTIONS:
Radiation: CyberKnife radiosurgery — Treatment Planning:
  Inverse planning using the CyberKnife planning system will be employed. The treatment plan used for each treatment will be based on an analysis of the volumetric dose including dose-volume histogram (DVH) analyses of the Planning Treatment Volume (PTV) and critical normal structures. The homogeneous CT model shall be used. Number of paths and beams used for each patient will vary and will be determined by the selected individual treatment plan. To reduce overall treatment time and total monitor units, 150-200 non-zero beams are recommended. No more than 250 beams shall be employed. Tuning structures shall be employed to minimize conformality index (CI) and new conformality index (nCI), preferably yielding values less than 1.20 and 1.25, respectively.

SUMMARY:
Radiation therapy is a well-established treatment modality for clinically localized prostate cancer. Men who choose to undergo radiation treatments for prostate cancer will have to live with the side effects for many years. Attempts have been made to protect surrounding tissues while delivering high dosage of radiation to cancer. With the rectum being so close to the prostate, many patients still suffer from side effects caused by radiation injury to the rectum, especially those who received conventional external beam radiotherapy.

CyberKnife is an FDA approved radiosurgical devise. Its flexible robotic arm allows radiation beams to be delivered in different directions, providing a highly conformal, uniform dose with steep dose gradients. Therefore, treatment with the CyberKnife radiosurgical system should minimize the toxicity to the surrounding structures. CyberKnife System also incorporates a dynamic tracking system to allow the robot to correct the targeting of therapeutic beams during treatment. These improvements allow for dose escalation within the prostate with less normal tissue toxicity.

The purpose of this study is to estimate the proportion of patients with endoscopically detectable telangiectasia as the indication of radiation injury to the rectum, after CyberKnife Treatment for prostate cancer.

DETAILED DESCRIPTION:
Radiation therapy is a well-established treatment modality for clinically localized prostate cancer. Current techniques include conventional external beam radiotherapy and intensity modulated radiation therapy (IMRT). The efficacy of conventional external beam radiation treatment (60-70 Gy in 2 Gy fractions) using several uniform fields has been documented. The 10-year disease-free survival rate for patients with disease confined to the prostate in the pre-Prostate Specific Antigen (PSA) era was approximately 50-70%. Analysis of these data suggested that dose escalation could improve local control in prostate cancer.

On average, men who choose to undergo radiation therapy treatments for prostate cancer will have to live with the side effects of therapy for many years. Chronic proctitis may occur after radiotherapy (RT) to the pelvic region. According to a published series, it clinically occurs after radiation therapy of localized prostate cancer at a frequency of 5-20%. It occurs months to years after treatment (average 8-12 months) with a large majority within two years following radiation therapy. Patient characteristics, such as a history of inflammatory bowel disease or chronic anticoagulation therapy, may increase an individual patient's risk of clinically significant proctitis. Patients with radiation-induced proctopathy have described symptoms of rectal pain, diarrhea, urgency, rectal bleeding, and increased frequency of bowel movements. Endoscopic evaluation shows telangiectasia, congested mucosa and ulcers. Rectal bleeding occurs from the neovascular telangiectasia seen in about 60% of patients receiving conventionally fractionated radiation therapy. The other symptoms probably develop from the decreased rectal compliance associated with rectal wall fibrosis. These symptoms are, in current reports, most often classified according to the NCI Common Toxicity Criteria grade for late gastrointestinal side effects. Due to the proximity of the rectum and bladder to the prostate, using conventional techniques, the prescription dose is limited to 65-70 Gy. Although attempts were made to protect the rectum, the incidence of rectal bleeding was unacceptable at doses greater than 70 Gy (20%).

The risk of proctitis and rectal bleeding appeared to be dependent upon both the radiation dose and the volume of the rectum in the high dose area. Radiation Oncologists' efforts to optimize the therapeutic ratio for prostate cancer treatment have therefore been directed toward limiting the high dose volume to the prostate while escalation the dose within that volume. Intensity modulated radiation therapy (IMRT) is a widely used technology to achieve this goal. It is accomplished by modulating the radiation beam intensity within each radiation field in accordance with an optimization algorithm. This has allowed greater dose-escalation without evident increase in acute complications, although follow-up is too short to fully assess control and complication rates. Whether IMRT will provide a degree of conformity that proves to eradicate prostate cancer with a high probability while sparing local structures is as yet unresolved.

Late Rectal Mucosal Injury Following CyberKnife RadioSurgery for Clinically Localized Prostate Cancer. The type, extent and incidence of rectal mucosal injury following CyberKnife radiosurgery are currently unknown. The severity of clinical proctitis following radiation therapy is commonly documented using the NCI Common toxicity criteria/Radiation Therapy Oncology Group/EORTC. Unfortunately, clinical proctitis has a low sensitivity for detecting rectal mucosal injury. Endoscopy gives the most accurate estimate of the extent and incidence of rectal mucosal injury. The Vienna rectoscopy score (VRS) was developed to quantify rectal mucosal changes following radiation therapy. In this study, endoscopic evaluation of mucosal damage from CyberKnife treatment will be documented and correlated with gastrointestinal side effects and treatment planning parameters.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate (Biopsy within one year of enrollment)
* Signed Study-Specific Consent
* PSA within 60 days of registration
* Baseline American Urological Association (AUA)/ International Prognostic Scoring System (IPSS) score of < 20
* Candidate for screening colonoscopy
* Pretreatment Colonoscopy/lower endoscopy done

Exclusion Criteria:

* Prior pelvic radiotherapy
* Prior radical prostate surgery
* Recent (within 5 years) or concurrent cancers other than non-melanoma skin cancer
* Implanted hardware adjacent to the prostate that would prohibit appropriate treatment planning and/or treatment delivery
* Inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Collins, MD,PhD, Principal Investigator — Georgetown University Hospital
Locations (1):
- MedStar Georgetown University Hospital, Washington, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CyberKnife Radiosurgery, Colonoscopy: CyberKnife radiosurgery for prostate cancer; bowel toxicity will be evaluated at 2 years by colonoscopy (lower endoscopy).
  CyberKnife radiosurgery: Treatment Planning:
  Inverse planning using the CyberKnife planning system will be employed. The treatment plan used for each treatment will be based on an analysis of the volumetric dose including dose-volume histogram (DVH) analyses of the PTV and critical normal structures. The homogeneous CT model shall be used. Number of paths and beams used for each patient will vary and will be determined by the selected individual treatment plan. To reduce overall treatment time and total monitor units, 150-200 non-zero beams are recommended. No more than 250 beams shall be employed. Tuning structures shall be employed to minimize conformality index (CI) and new conformality index (nCI), preferably yielding values less than 1.20 and 1.25, respectively.
Period: Overall Study
Arm/Group | CyberKnife Radiosurgery, Colonoscopy
Started | 4
Completed | 0
Not Completed | 4
Not completed — slow accrual, trial closed prematurely. | 4

BASELINE CHARACTERISTICS:
Arm/Group | CyberKnife Radiosurgery, Colonoscopy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 75.5 [74 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Endoscopically Detectable-telangiectasia (VRS Grade 1 or Higher).
Description: Telangiectasia is the primary outcome since it is a measure of tissue fibrosis (primary source of proctitis) and is a well-defined and measurable outcome.
  No patients had outcome before the trial was terminated.
Time Frame: Planned for 7 years, collected up to 23 months
Measure: Count of Participants; unit: Participants
Arm/Group | CyberKnife Radiosurgery, Colonoscopy
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Proportion of Patients With Rectal Bleeding.
Time Frame: Planned for 7 years, collected up to 23 months
Population: No patients had outcome before the trial was terminated.
Measure: Count of Participants; unit: Participants
Groups:
- CyberKnife Radiosurgery, Colonoscopy: CyberKnife radiosurgery for prostate cancer; bowel toxicity will be evaluated at 2 years by colonoscopy (lower endoscopy).
  CyberKnife radiosurgery: Treatment Planning:
  Inverse planning using the CyberKnife planning system will be employed. The treatment plan used for each treatment will be based on an analysis of the volumetric dose including dose-volume histogram (DVH) analyses of the Planning Treatment Volume (PTV) and critical normal structures. The homogeneous CT model shall be used. Number of paths and beams used for each patient will vary and will be determined by the selected individual treatment plan. To reduce overall treatment time and total monitor units, 150-200 non-zero beams are recommended. No more than 250 beams shall be employed. Tuning structures shall be employed to minimize conformality index (CI) and new conformality index (nCI), preferably yielding values less than 1.20 and 1.25, respectively.
Arm/Group | CyberKnife Radiosurgery, Colonoscopy
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be defined as the time in months from study entry until progression or death. Patients who are alive and free from progression on the date of closing follow-up will be censored on that date. Data table reports the number of participants who were alive without progression at the end of the study.
Time Frame: Planned for 7 years, collected up to 23 months
Measure: Count of Participants; unit: Participants
Arm/Group | CyberKnife Radiosurgery, Colonoscopy
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: This study was open for accrual for 23 months total. This study was closed due to low accrual.
Description: A total of 4 subjects out of 40 were accrued for this study. None of the 4 subjects have experienced any adverse events since the start of this study.
Arm/Group | CyberKnife Radiosurgery, Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No